CLINICAL TRIAL: NCT02227914
Title: Phase 1b/2 Study of Oprozomib in Combination With Sorafenib in Subjects With Advanced Hepatocellular Carcinoma
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Study stopped due to administrative reasons
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OPZ011; 2014-003149-85 (EudraCT Number)
Record Dates: First submitted 2014-08-26; First posted 2014-08-28 (Estimated); Last update posted 2017-05-02 (Actual); Status verified 2017-04

CONDITIONS: Advanced Hepatocellular Carcinoma
MeSH Terms: interventions — ONX 0912; Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Oprozomib with Sorafenib (Experimental): Phase 1b:
  Oprozomib doses will be escalated in sequential groups of at least 2 subjects. Study subjects will receive oprozomib at dose levels of 90, 120, 150, 180, 210, or 240 mg + sorafenib to reach the dose levels of 600 or 800 mg total daily dose until the maximum tolerated dose (MTD) is reached.
  Phase 2:
  Study subjects who meet the entry criteria will receive oprozomib + sorafenib at the RP2D (recommended Phase 2 dose) established in the Phase 1b portion of the study.
  Interventions: Drug: Oprozomib; Drug: Sorafenib
- Sorafenib (Active Comparator): Phase 2:
  Study subjects who meet the entry criteria will receive sorafenib 400 mg twice a day (800 mg total daily dose).
  Interventions: Drug: Sorafenib

INTERVENTIONS:
Drug: Oprozomib — Study subjects will receive oprozomib tablets once a day on Days 1, 2, 8, 9, 15, 16, 22 and 23 of a 28 day cycle
  Arms: Oprozomib with Sorafenib
Drug: Sorafenib — Study subjects will receive sorafenib tablets twice a day for Days 1-28

SUMMARY:
The purpose of Phase 1b of the study is to determine the maximum tolerated dose, pharmacokinetics (PK) and pharmacodynamics (PDn) and assess the safety, tolerability and activity of oprozomib in combination with sorafenib in subjects with advanced hepatocellular carcinoma (HCC).

The purpose of Phase 2 of the study is to evaluate the efficacy of oprozomib in combination with sorafenib versus sorafenib alone and to compare the key outcome measures for subjects with advanced HCC.

ELIGIBILITY:
Key Inclusion Criteria:

1. Patients with advanced HCC
2. For the Phase 2 portion of the study, at least 1 measurable tumor lesion according to Response Evaluation Criteria in Solid Tumors (RECIST) 1.1, which has not been previously treated with local therapy
3. Cirrhotic status of Child-Pugh Class A only
4. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1
5. The following laboratory parameters:

   * Albumin ≥ 2.8 g/dL
   * Platelet count ≥ 60,000/mm3
   * Absolute neutrophil count (ANC) ≥ 1500/mm3
   * Hemoglobin ≥ 8.5 g/dL
   * Total bilirubin ≤ 3 mg/dL
   * Alanine aminotransaminase (ALT) and aspartate aminotransferase (AST) ≤ 3 times upper limit of normal (ULN)
   * Amylase and lipase ≤ 1.5 times ULN
   * Calculated or measured creatinine clearance (CrCl) ≥ 30 mL/min
   * Prothrombin time (PT)-international normalized ratio (INR) ≤ 2.3 or PT ≤ 6 seconds above control

Key Exclusion Criteria:

1. Previous or concurrent cancer that is distinct in primary site or histology from HCC, EXCEPT cervical and breast carcinoma in situ, adequately treated basal cell or squamous cell carcinoma of the skin, or superficial bladder tumors (Ta, Tis & T1)
2. Renal failure requiring hemo- or peritoneal dialysis
3. History of cardiac disease
4. Active clinically serious infections. Hepatitis B is allowed if no active replication is present. Hepatitis C is allowed if no antiviral treatment is required
5. Known history of human immunodeficiency virus (HIV) infection
6. Known history or symptomatic metastatic brain or meningeal tumors
7. Clinically significant gastrointestinal (GI) bleeding, serious nonhealing wound and ulcer within 3 months prior to study entry, or bone fracture within 30 days prior to study entry
8. History of organ allograft
9. Known or suspected allergy to the investigational agent or any agent given in association with this trial
10. Inability to swallow medication, inability or unwillingness to comply with the drug administration requirements, or GI condition that could interfere with the oral absorption or tolerance of treatment
11. Uncontrolled diabetes
12. Any contraindication to oral hydration (e.g., preexisting cardiac impairment or fluid restriction)
13. Uncontrolled ascites
14. Pleural effusion or ascites that causes respiratory compromise (NCI-CTCAE ≥ Grade 2 dyspnea).
15. Women who are pregnant and/or breastfeeding
16. Prior use of any systemic anticancer chemotherapy for HCC
17. Prior use of systemic investigational agents for HCC
18. Concomitant treatment with strong cytochrome P450 3A4 (CYP3A4) inhibitors
19. Known hypersensitivity or intolerance to dexamethasone or 5-HT3 antagonist

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-12; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) - Phase 1b | 16 months
  To determine the maximum tolerated dose (MTD) and identify the recommended Phase 2 dose (RP2D) of oprozomib in combination with sorafenib in subjects with advanced hepatocellular carcinoma (HCC).
Time To Progression (TTP) - Phase 2 | 16 months
  To evaluate the efficacy of oprozomib in combination with sorafenib versus sorafenib alone in subjects with advanced HCC, as measured by time to progression (TTP), defined as time from randomization to disease progression.

SECONDARY OUTCOMES:
Adverse Events (AEs) and Serious Adverse Events (SAEs) - Phase 1b & Phase 2 | Until 30 days after the end of study (32 months)
  Number of patients that experience Adverse Events (AEs). Adverse Events (AEs) and Serious Adverse Events (SAEs) graded according to the NCI-CTCAE (Version 4.03).
Pharmacokinetics (PK) parameters - Phase 1b | 16 months
  Evaluate population pharmacokinetic (PK) parameters, including maximum plasma concentration (Cmax), time to maximum plasma concentration (Tmax), area under the curve at the last measurable time point (AUC0-t), and area under the curve extrapolated to infinity (AUC0-inf) using noncompartmental methods.
Pharmacodynamic (PDn) parameter - Phase 1b | 16 months
  The extent of inactivation of proteasome activity in red blood cells (RBCs) after oprozomib dosing will be monitored as a PDn parameter. Pharmacodynamic inhibition will be listed by dose cohort, exposure, and response status.
Overall Response Rate (ORR) - Phase 2 | 16 months
  To estimate the overall response rate (ORR), defined as the proportion of subjects with a best overall response of complete response (CR) and partial response (PR) for subjects receiving oprozomib in combination with sorafenib and for subjects receiving sorafenib alone.
Progression-free Survival (PFS) - Phase 2 | 16 months
  Progression-free survival (PFS), defined as time from randomization to the earlier of PD or death due to any cause.
Overall Survival (OS) - Phase 2 | 16 months
  Overall survival (OS) is defined as time from randomization to death due to any cause.

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (6):
- United States (6):
  - Lahey Hospital & Medical Center, Burlington, California
  - Rocky Mountain Cancer Centers, Denver, Colorado
  - University of Miami Hospital & Clinics, Miami, Florida
  - The University of Chicago Medical Center, Chicago, Illinois
  - The Ohio State University, Martha Morehouse Medical Plaza, Columbus, Ohio
  - University of Wisconsin Comprehensive Cancer Center, Madison, Wisconsin